CLINICAL TRIAL: NCT06063317
Title: A Phase I, Dose Escalation and Dose Expansion, Safety and Tolerability Study of onCARlytics (CF33-CD19), Administered Intravenously or Intratumorally in Combination With Blinatumomab in Adults With Advanced or Metastatic Solid Tumors (OASIS)
Brief Title: A Study of onCARlytics (CF33-CD19) in Combination With Blinatumomab in Adults With Advanced or Metastatic Solid Tumors (OASIS)
Acronym: OASIS
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Imugene Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF33-CD19-101
Record Dates: First submitted 2023-09-14; First posted 2023-10-02 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult
Keywords: Immunotherapy; Oncolytic Virus; Bispecific T-Cell Engager; BiTE; Blincyto
MeSH Terms: conditions — Bites and Stings | interventions — blinatumomab; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CF33-CD19 IT Administration Monotherapy (Experimental)
  Interventions: Biological: CF33-CD19 IT Monotherapy
- CF33-CD19 IV Administration Monotherapy (Experimental)
  Interventions: Biological: CF33-CD19 IV Monotherapy
- CF33-CD19 IT Administration in Combination with Blinatumomab (Experimental)
  Interventions: Biological: CF33-CD19 IT Combination; Drug: Blinatumomab
- CF33-CD19 IV Administration in Combination with Blinatumomab (Experimental)
  Interventions: Biological: CF33-CD19 IV Combination; Drug: Blinatumomab
- CF33-CD19 IT Administration in Combination with Blinatumomab and Hydroxyurea (Experimental)
  Interventions: Biological: CF33-CD19 IT Combination; Drug: Blinatumomab; Drug: Hydroxyurea
- CF33-CD19 IV Administration in Combination with Blinatumomab and Hydroxyurea (Experimental)
  Interventions: Biological: CF33-CD19 IV Combination; Drug: Blinatumomab; Drug: Hydroxyurea

INTERVENTIONS:
Biological: CF33-CD19 IT Monotherapy — Safety Run-In Phase: CF33-CD19 will be administered intratumorally on Days 1 and 8 of Cycle 1 and Day 1 of each subsequent 21-day cycle.
  Arms: CF33-CD19 IT Administration Monotherapy
Biological: CF33-CD19 IV Monotherapy — Safety Run-In Phase: CF33-CD19 will be administered intravenously on Days 1 and 8 of Cycle 1 and Day 1 of each subsequent 21-day cycle.
  Arms: CF33-CD19 IV Administration Monotherapy
Biological: CF33-CD19 IT Combination — Dose Escalation Combination Phase: CF33-CD19 will be administered intratumorally on Days 1 and 15 of each 28 day cycle.
  Arms: CF33-CD19 IT Administration in Combination with Blinatumomab; CF33-CD19 IT Administration in Combination with Blinatumomab and Hydroxyurea
Biological: CF33-CD19 IV Combination — Dose Escalation Combination Phase: CF33-CD19 will be administered intravenously on Days 1 and 15 of each 28 day cycle.
  Arms: CF33-CD19 IV Administration in Combination with Blinatumomab; CF33-CD19 IV Administration in Combination with Blinatumomab and Hydroxyurea
Drug: Blinatumomab — Blinatumomab will be infused via a 7-day continuous infusion from Days 2-9 and Days 16-23 of each 28-day cycle.
  Arms: CF33-CD19 IT Administration in Combination with Blinatumomab; CF33-CD19 IT Administration in Combination with Blinatumomab and Hydroxyurea; CF33-CD19 IV Administration in Combination with Blinatumomab; CF33-CD19 IV Administration in Combination with Blinatumomab and Hydroxyurea
Drug: Hydroxyurea — Hydroxyurea will be orally administered daily.
  Arms: CF33-CD19 IT Administration in Combination with Blinatumomab and Hydroxyurea; CF33-CD19 IV Administration in Combination with Blinatumomab and Hydroxyurea

SUMMARY:
This is an open-label, dose escalation and dose expansion, multi-center phase I study evaluating the safety and tolerability of CF33-CD19 administered intravenously (IV) or intratumorally (IT) in combination with blinatumomab and with or without hydroxyurea in adults with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
CF33-CD19, a novel chimeric orthopoxvirus, will be administered as a monotherapy or in combination with blinatumomab and with or without hydroxyurea to assess the safety and efficacy of the treatment regimens as well as immunological changes in the tumour microenvironment.

Subjects eligible for treatment include those with any metastatic or advanced solid tumor who have documented radiological progression per RECIST following at least two prior lines of therapy.

All enrolled monotherapy subjects will be treated with CF33-CD19 on Day 1 and 8 of Cycle 1 and then on Day 1 of each 21-day cycle thereafter. Subjects treated with the combination regimen will receive CF33-CD19 on Days 1 and 15 of each 28-day cycle. In addition, they will receive blinatumomab as a 7-day continuous infusion from Days 2-9 and Days 16-23 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from subject or legally authorized representative.
2. Age ≥ 18 years old on the date of consent.
3. Life expectancy of at least 3 months.
4. Any histologically or cytologically confirmed advanced or metastatic solid tumor with documented radiological progression per RECIST v1.1. Eligible subjects must have received at least two prior lines of approved therapies, including targeted therapies, for which they are eligible and failed or relapsed on or after that treatment.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1.
6. At least one measurable lesion as defined by RECIST v1.1 criteria.
7. Adequate renal function.
8. Adequate hepatic function.
9. Adequate hematologic function.
10. Willing and able to comply with scheduled visits, study treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Prior treatment with a poxvirus based oncolytic virus or a bispecific CD19-directed CD3 T-cell engager.
2. Continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 4 weeks prior to first dose of study treatment.
3. Any radiation within 2 weeks of start of study treatment.
4. Active autoimmune disease.
5. Current or history of severe skin disease with open wounds.
6. History of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease.
7. History of pancreatitis.
8. Prior allogeneic tissue/organ transplant or other medical conditions requiring ongoing treatment with immunosuppressive drugs or any condition resulting in a systemic immunosuppressed state.
9. Medical history of central nervous system (CNS) metastases unless the subject has completed definitive treatment for the CNS lesions with whole brain radiation therapy (WBRT) or stereotactic radiosurgery (SRS) and are neurologically stable, asymptomatic, and off corticosteroids for at least 2 months prior to first dose.
10. History of documented congestive heart failure (New York Heart Association [NYHA] class II - IV), unstable angina, poorly controlled hypertension, clinically significant valvular heart disease or high-risk uncontrolled arrhythmias.
11. Bleeding diathesis due to underlying medical condition or ongoing anticoagulation medication.
12. History or presence of clinically relevant CNS pathology, or any other CNS disability judged by the Investigator to be clinically significant and precluding informed consent or participation in the study.
13. Active infection requiring systemic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
All Treatment Arms - Incidence and severity of Adverse Events | From first dose of study drug through 30 days following the last dose of study treatment
  Adverse events will be graded according to CTCAE v5.0.
Monotherapy Treatment Arms - Determination of the Recommended Phase 2 Dose (RP2D) to apply to Dose Escalation Combination Phase as supported by immune response as seen in lymphocyte subsets | From first dose of study drug through treatment discontinuation, an average of 6 months
  Change in lymphocyte subset expression in tumor tissue and peripheral blood pre and post dose
Monotherapy Treatment Arms - Determination of RP2D to apply to Dose Escalation Combination Phase as supported by immune response as seen in cytokines | From first dose of study drug through treatment discontinuation, an average of 6 months
  Change in cytokine levels in peripheral blood pre and post dose
Monotherapy Treatment Arms - Determination of RP2D to apply to Dose Escalation Combination Phase as supported by anti-tumor activity | From first dose of study drug through treatment discontinuation, an average of 6 months
  Stable Disease and Response (PR and CR) based on RECIST v1.1 and iRECIST v1.0.

SECONDARY OUTCOMES:
Combination Treatment Arms - Determination of the Recommended Phase 2 Dose (RP2D) for CF33-CD19 + blinatumomab + hydroxyurea combination as supported by immune response as seen in lymphocyte subsets | From first dose of study drug through treatment discontinuation, an average of 6 months
  Change in lymphocyte subset expression in tumor tissue and peripheral blood pre and post dose
Combination Treatment Arms - Determination of RP2D for CF33-CD19 + blinatumomab + hydroxyurea combination as supported by immune response as seen in cytokines | From first dose of study drug through treatment discontinuation, an average of 6 months
  Change in cytokine levels in peripheral blood pre and post dose
Combination Treatment Arms - Determination of RP2D for CF33-CD19 + blinatumomab + hydroxyurea combination as supported by anti-tumor activity | From first dose of study drug through treatment discontinuation, an average of 6 months
  Stable Disease and Response (PR and CR) based on RECIST v1.1 and iRECIST v1.0.
All Treatment Arms - Overall Response Rate | From first dose of study drug through treatment discontinuation, an average of 6 months
  Overall Response Rate (ORR) is defined as the proportion of subjects in the efficacy population who achieve a radiographic Investigator-assessed confirmed CR or PR, per RECIST v1.1 or confirmed iCR or iPR per iRECIST v1.0.
All Treatment Arms - Progression Free Survival | From first dose of study drug through treatment discontinuation, an average of 6 months
  Progression Free Survival (PFS) defined as the time from first dose of study drug to first documentation of PD based on RECIST 1.1, or to death from any cause.
All Treatment Arms - Duration of Response | From first dose of study drug through treatment discontinuation, an average of 6 months
  Duration of Response (DoR) measured as the time from the date a response of PR/iPR or better was first recorded to the date on which progressive disease was first noted or the date of death due to any cause.
All Treatment Arms - Disease Control Rate | From first dose of study drug through treatment discontinuation, an average of 6 months
  Disease Control Rate (DCR), measured as the proportion of subjects who achieve an Investigator-assessed confirmed CR/iCR, PR/iPR, or Stable Disease (SD)/immune SD (iSD) per RECIST v1.1 and iRECIST v1.0.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Northwestern, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Imugene Limited (ASX: IMU) is a publicly-listed Australian biotechnology company developing cancer immunotherapies. — http://www.imugene.com/